CLINICAL TRIAL: NCT05600322
Title: A Prospective, Comparative Within Patient Controlled, Multi-center Study of Hexvix Blue Light Cystoscopy and White Light Cystoscopy in the Detection of Bladder Cancer
Brief Title: Comparative Study of Hexvix Blue Light Cystoscopy and White Light Cystoscopy in the Detection of Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Photocure (Industry)
Collaborators: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry); Richard Wolf GmbH (Industry); Tigermed-Jyton Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PC B309/21 / YHCT-HEX-B1
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: This is a prospective, comparative, within patient controlled, multi-center study of Hexvix Blue light cystoscopy and standard White light cystoscopy in the detection of bladder cancer. Patients with suspicious or confirmed bladder cancer will be enrolled and there will be a maximum of three regular study visits for each patient. Visit 1 is a screening visit, Visit 2 is the cystoscopic examinations and Visit 3 is the safety follow-up.
  At Visit 2, enrolled patients will be instilled with 50 mL Hexvix solution in the bladder for one hour. After bladder evacuation, the inspection of the bladder and mapping of lesions seen under White light will be done. Secondly, inspection of the bladder and mapping of lesions seen under Blue light will be done. The Richard Wold PDD system (System Blue) will be used. Lesions detected will be resected or biopsied and sent to the local and central pathologists for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hexvix Blue light cystoscopy (Experimental): In this study, enrolled patients will undergo standard White light cystoscopy and Blue light cystoscopy following Hexvix administration. Lesions detected during the cystoscopies will be resected or biopsied.
  Interventions: Drug: Hexaminolevulinate Hydrochloride; Device: Richard Wolf Photodynamic Diagnostic Equipment (PDD) system

INTERVENTIONS:
Drug: Hexaminolevulinate Hydrochloride — Enrolled patients will be instilled with 50 mL hexaminolevulinate hydrochloride as intravesical solution (Hexvix) in the bladder for one hour at Visit 2. After bladder evacuation, the cystoscopic examinations will be performed in both white and blue light.
  Other Names: Hexvix
Device: Richard Wolf Photodynamic Diagnostic Equipment (PDD) system — Cystoscopy in White and Blue light will be done using the Richard Wolf PDD system.
  Other Names: System Blue

SUMMARY:
A study to compare Hexvix Blue light cstoscopy with standard White light cystoscopy in the detection of bladder cancer.

DETAILED DESCRIPTION:
A phase III, prospective, within patient controlled, multi-center study to compare Blue light cystoscopy with Hexvix and standard White light cystoscopy in the detection of bladder cancer, to evaluate the efficacy and safety of Hexvix Blue light cystoscopy in Chinese population.

Patients with suspicious or confirmed bladder cancer will participate in the trial and undergo Blue light cystoscopy with Hexvix in addition to the standard White light cystoscopy. Specific clinical questions will be asked:

* What is the proportion of patients who have at least one specific kind of tumor found by Blue light cystoscopy with Hexvix but not by White light cystoscopy?
* What is the proportion of patients who have at least one specific kind of lesion found by Blue light cystoscopy with Hexvix but not by White light cystoscopy?
* What is the proportion of false positive lesions detected with Hexvix Blue light cystoscopy and White light cystoscopy?
* What is the proportion of patients with Adverse Events (AE) during the study?

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical study; thoroughly informed, signed and dated the informed consent form; willing to follow and have the ability to complete all trial procedures.
2. Suspicious or confirmed patients with bladder cancer.
3. Age 18 or older.

Exclusion Criteria:

1. Gross haematuria. (Note: Gross haematuria is defined as a heavy bladder bleed resulting in marked amounts of blood in the urine, which may visually limit cystoscopy. Where the haematuria is light, the patient should not be excluded, if in the investigator's opinion, rinsing and/or electro-cautery during cystoscopy will alleviate the possible interference with cystoscopy).
2. Patients who have received BCG immunotherapy or intravesical chemotherapy within the past 6 weeks prior to the procedure.
3. Porphyria.
4. Known allergy to hexaminolevulinate hydrochloride or a similar compound.
5. Pregnancy or breast-feeding or women who plan to become pregnant during the trial, and men or women who are unwilling to take barrier contraceptives from 2 weeks before application of investigational medication to 28 days after application of investigational medication (Note: All women of child-bearing potential must document a negative urine pregnancy test before study inclusion and use adequate contraception during the study.
6. Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days.
7. Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
8. Patients that the investigator assessed unsuitable to the study.
9. Subjects with contraindications to white light cystoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Han Zhong, BMed, Principal Investigator — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangzhou Province
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin City

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hexvix Blue Light Cystoscopy
Started | 158
Completed | 157
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: In the group of 158 enrolled subjects, 37 subjects were training patients. To reduce possible bias in the assessment of the objectives, 6 subjects were randomized to not continue with blue light cystoscopy. In addition, 1 patient withdrew. Baseline characteristics are reported for the 114 subjects that underwent both white and blue light cystoscopy.
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han nationality | 112
  Others | 2
Region of Enrollment [Number; unit: participants]
  China | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Histology-confirmed Lesions (Ta, T1, or CIS) Who Have at Least One Such Lesion Found by Hexvix Blue Light Cystoscopy But Not by White Light Cystoscopy.
Description: In the subsection of patients with histology-confirmed lesions (Ta, T1, or CIS) , the number of patients who have at least one such lesion found by Hexvix blue light cystoscopy but not by white light cystoscopy is measured.
Time Frame: 1 day (At time of cystoscopy examination)
Population: Patients with histology-confirmed lesions (Ta, T1, or CIS) were included in the Modified Full Analysis Set (mFAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 97
Participants | 42

2. Secondary Outcome: Number of Subjects With at Least One Additional CIS Lesion Detected With Hexvix Blue Light Cystoscopy But Not With White Light Cystoscopy.
Time Frame: 1 day (At time of cystoscopy examination)
Population: Patients randomised to undergo white light cystoscopy and Hexvix blue light cystoscopy were included in the Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 114
Participants | 11

3. Secondary Outcome: Number of Lesions Detected With Hexvix Blue Light Cystoscopy and White Light Cystoscopy for Following Lesion Types (Papillary Urothelial Neoplasm of Low Malignant Potential (PUNLMP), Carcinoma in Situ (CIS), Ta, T1, T2-T4).
Time Frame: 1 day (At time of cystoscopy examination)
Population: The total number of lesions in the full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 114
Number analyzed (Lesions) | 306
percentage of lesions
  PUNLMP lesion detection rate Blue light | 0 [NA to NA] — 0 PUNLMP lesions detected in Blue light
  PUNLMP lesion detection rate White light | 0 [NA to NA] — 0 PUNLMP lesions detected in Blue light
  CIS lesion detection rate Blue light | 94.7 [74.0 to 99.9]
  CIS lesion detection rate White light | 42.1 [20.3 to 66.5]
  Ta lesion detection rate Blue light | 100 [98.4 to 100]
  Ta lesion detection rate White light | 76.1 [70.0 to 81.5]
  T1 lesion detection rate Blue light | 98.2 [90.6 to 100]
  T1 lesion detection rate White light | 91.2 [80.7 to 97.1]
  T2-T4 lesion detection rate Blue light | 100 [39.8 to 100]
  T2-T4 lesion detection rate White light | 100 [39.8 to 100]

4. Secondary Outcome: The Proportion of False Positive Lesions Detected With Hexvix Blue Light Cystoscopy and White Light Cystoscopy.
Time Frame: 1 day (At time of cystoscopy examination)
Population: Patients that were randomised to undergo standard White light cystoscopy and Hexvix Blue light cystoscopy.
Measure: Number (95% Confidence Interval); unit: percentage of false positive lesions
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 114
percentage of false positive lesions
  False positive detection rate Blue light | 23.2 [19.2 to 27.7]
  False positive detection rate White light | 16.0 [11.9 to 20.8]

5. Other Pre Specified Outcome: The Number of Patients With Adverse Events (AE) During the Study.
Time Frame: 1 week
Population: Patients who received Hexvix instillation were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Hexvix Blue Light Cystoscopy
Number analyzed (Participants) | 158
Participants | 95

ADVERSE EVENTS:
Time Frame: Approx. 3 weeks, including time from screening visit (- 2 weeks) until safety follow-up of 1 week.
Arm/Group | Hexvix Blue Light Cystoscopy
All-Cause Mortality (participants affected / at risk) | 0/158
Serious Adverse Events (participants affected / at risk) | 0/158
Other Adverse Events (participants affected / at risk) | 95/158
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hexvix Blue Light Cystoscopy (N=158)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 10
Dysuria (Renal and urinary disorders) | 6
Urethral pain (Renal and urinary disorders) | 6
Bladder spasm (Renal and urinary disorders) | 3
Bladder pain (Renal and urinary disorders) | 2
Ureteral spasm (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Urethral syndrome (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary tract spasm (Renal and urinary disorders) | 1
Blood bilirubin increased (Investigations) | 14
Blood pressure increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Blood albumin decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
Incision site pain (Injury, poisoning and procedural complications) | 17
Post procedural haematuria (Injury, poisoning and procedural complications) | 2
Constipation (Gastrointestinal disorders) | 9
Abdominal pain lower (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 2
Dyschezia (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 13
Pyrexia (General disorders) | 6
Fatigue (General disorders) | 1
Inflammation (General disorders) | 1
Peripheral swelling (General disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vitreous floaters (Eye disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT05600322/Prot_SAP_000.pdf